CLINICAL TRIAL: NCT03035331
Title: Phase I/II Study of Dendritic Cell Therapy Delivered Intratumorally After Cryoablation and Anti-PD-1 Antibody (Pembrolizumab) for Patients With Non-Hodgkin Lymphoma
Brief Title: Dendritic Cell Therapy, Cryosurgery, and Pembrolizumab in Treating Patients With Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1685; NCI-2017-00113 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1685 (Other: Mayo Clinic in Rochester); P50CA097274 (NIH); 16-005856 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-12

CONDITIONS: Aggressive Non-Hodgkin Lymphoma; Indolent Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cryosurgery; pembrolizumab; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, dendritic cell therapy, cryosurgery) (Experimental): Patients receive pembrolizumab IV on day 1. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive dendritic cell therapy IT on days 2, 8, and 15 of cycles 2 and 3, and day 2 of cycles 4 and 5. Patients undergo cryosurgery on day 2 of cycle 2 and receive pneumococcal 13-valent conjugate vaccine by injection on day 2 of cycles 2-5. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients who are CR, PR, or SD after completion of therapy, may receive pembrolizumab for an additional 18 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Cryosurgery; Biological: Dendritic Cell Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Biological: Pneumococcal 13-valent Conjugate Vaccine; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Cryosurgery — Undergo cryosurgery
  Other Names: Ablation, Cryo; Cryoablation; cryosurgical ablation
Biological: Dendritic Cell Therapy — Given IT
  Other Names: Dendritic Cell Vaccine Therapy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Pneumococcal 13-valent Conjugate Vaccine — Given by injection
  Other Names: PCV 13; PCV13 Vaccine; Prevnar 13
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I/II trial studies the best dose and side effects of dendritic cell therapy, cryosurgery and pembrolizumab in treating patients with non-Hodgkin lymphoma. Vaccines, such as dendritic cell therapy made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells. Cryosurgery kills cancer cells by freezing them. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving dendritic cell therapy, cryosurgery and pembrolizumab may work better at treating non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the optimal dose schedule, safety and tolerability as measured by the incidence of significant toxicity of combination therapy with anti-PD-1 monoclonal antibody, cryoablation, and intra-tumor injection of autologous dendritic cell into the cryoablated tumor. (Phase I) II. Test the efficacy (overall response rate) of combination therapy with anti-PD-1 monoclonal antibody, cryoablation, and intra-tumor injection of autologous dendritic cell vaccine. (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate the feasibility of this combination immunotherapy. (Phase I) II. Evaluate patient quality of life. (Phase I) III. Evaluate the partial response (PR) and complete response (CR) rate of this combination immunotherapy. (Phase II) IV. Evaluate the progression free survival, treatment free survival, duration of response, disease-free rate at 2 years, and overall survival of this combination immunotherapy. (Phase II) V. Evaluate the safety of this combination immunotherapy. (Phase II)

CORRELATIVE OBJECTIVES:

I. Assess the effect of combination immunotherapy on patients' immune status and anti-tumor immune response. (Phase II) II. Assess the potential association between PD-1/PD-L1/PD-L2 expression in tumor and blood with clinical efficacy. (Phase II) III. Assess the potential association between tumor antigen mutations and antigen-specific immune response with clinical efficacy. (Phase II) IV. Evaluate patient quality of life. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive pembrolizumab intravenously (IV) on day 1. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive dendritic cell therapy intratumorally (IT) on days 2, 8, and 15 of cycles 2 and 3, and day 2 of cycles 4 and 5. Patients undergo cryosurgery on day 2 of cycle 2 and receive pneumococcal 13-valent conjugate vaccine by injection on day 2 of cycles 2-5. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients who are CR, PR, or stable disease (SD) after completion of therapy, may receive pembrolizumab for an additional 18 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months during the first year post-treatment, every 4 months during the second year post-treatment, and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of biopsy-proven non-Hodgkin lymphoma, excluding chronic lymphocytic leukemia, primary central nervous system (CNS) lymphoma and Burkitt's lymphoma; Note: small lymphocytic lymphoma (SLL) is allowed
* Patients with indolent non-Hodgkin lymphoma (NHL) must have had >= 1 regimen of rituximab-containing regimen; Note: this includes follicular lymphoma (FL), marginal lymphoma and mucosa-associated lymphoid tissue (MALT)
* Patients with aggressive NHL must have had >= 2 regimens; Note: This includes diffuse large B cell lymphoma (DLBCL), mantle cell lymphoma (MCL), primary mediastinal large B-cell lymphoma (PMBCL), and T cell lymphoma
* Patient with aggressive NHL must have received prior therapy - at a minimum:

  * Anti-CD20 monoclonal antibody unless tumor is CD20 negative and
  * An anthracycline containing regimen
  * Transformed FL must have had therapy for FL and be refractory to chemotherapy for DLBCL
* Chemotherapy refractory disease in aggressive NHL is defined as

  * Stable disease of =< 12 months or progressive disease as best response to most recent chemotherapy containing regimen
  * Disease progression or recurrence =< 12 months of prior autologous stem cell transplantation (SCT)
* Patients with aggressive NHL must have failed autologous hematopoietic stem cell transplantation (HSCT), or are ineligible or not consenting to autologous HSCT
* Patient must have at least 3 measurable lesions that are >= 1.5 cm in one dimension; one of the lesions must be >= 2.0 cm and is amenable to image-guided cryoablation and multiple vaccine injections as determined by interventional radiology and principal investigator (PI) (including tumors that can be safely accessed using imaging guidance and treated with minimal risk to adjacent structures)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Absolute lymphocyte count >= 200/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 50,000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert's disease (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST/serum glutamic-oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Creatinine =< 1.5 x ULN or calculated creatinine clearance >= 60 mL/min for subject with creatinine ˃ 1.5 x institutional ULN (obtained =< 14 days prior to registration)
* Negative serum pregnancy test for women of childbearing potential =< 7 days prior to registration; Note: a second pregnancy test may be required =< 72 hours prior to receiving the first dose of study medication
* Negative human immunodeficiency virus (HIV), hepatitis B and C, and tuberculosis (TB) test
* Provide written informed consent
* Willing to return to the enrolling institution for follow-up (during active treatment and active monitoring phase of the study)
* Ability to complete questionnaire(s) by themselves or with assistance
* Willing to provide tissue and blood samples for research purposes
* Willing to use adequate contraception while on the study and until 120 days after the last dose of study drug

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Serious non-malignant disease such as active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations or other conditions which in the opinion of the investigator would compromise protocol objectives
* Currently receiving or have received any other investigational agent considered as a treatment for the primary neoplasm =< 28 days or within 4 half-lives (whichever is shorter) of the agent prior to registration
* History of other primary malignancy requiring systemic treatment within 6 months of protocol enrollment; patients must not be receiving chemotherapy or immunotherapy for another cancer; patients must not have another active malignancy requiring active treatment with the following acceptable EXCEPTIONS:

  * Basal cell carcinoma, squamous cell carcinoma, or melanoma of the skin that has undergone or will undergo potentially curative therapy
  * In situ cervical cancer that has undergone or will undergo potentially curative therapy
* Prior allogeneic bone marrow or peripheral blood stem cell transplantation
* Prior autologous bone marrow or peripheral blood stem cell transplantation =< 100 days prior to registration or if recovery from the transplant is inadequate
* Major surgery other than diagnostic surgery =< 4 weeks prior to registration
* Prior chemotherapy or radiation therapy =< 2 weeks prior to registration or who has not recovered (i.e. to =< grade 1 or baseline) from an adverse event due to the previously administered therapy
* History of hypersensitivity and anaphylactoid reactions to pneumococcal vaccine or any component of the formulation, including diphtheria toxoid
* Active autoimmune disease such as Crohn's disease, rheumatoid arthritis, Sjogren's disease, systemic lupus erythematosus, or similar conditions requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease/syndrome difficult to control in the past

  * EXCEPTIONS:

    * Vitiligo or resolved childhood asthma/atopy
    * Intermittent use of bronchodilators or local steroid injections
    * Hypothyroidism stable on hormone replacement,
    * Diabetes stable with current management
    * History of positive Coombs test but no evidence of hemolysis
    * Psoriasis not requiring systemic treatment
    * Conditions not expected to recur in the absence of an external trigger
* Coagulopathy, including the use of Coumadin or heparin anticoagulants that cannot be discontinued for the cryoablation procedure; NOTE: heparin for line patency without detectable lab abnormalities for coagulation will be allowed
* Corticosteroid use =< 2 weeks prior to registration; NOTE: patients must be off corticosteroids for at least 2 weeks prior to registration; this includes oral, IV, subcutaneous, or inhaled route of administration; patients on chronic corticosteroid for adrenal insufficiency or other reasons may enroll if they receive less than 10 mg/day of prednisone (or equivalent)
* Active CNS malignancy
* Evidence of interstitial lung disease or active, non-infectious pneumonitis
* Received a live vaccine =< 30 days prior to registration
* New York Heart Association classification III or IV cardiovascular disease or recent myocardial infarction or unstable angina pectoris or cardiac arrhythmia =< 30 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lin, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1; Phase 2 Dose Level 1: Patients receive 200mg pembrolizumab IV on day 1. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive an injection of between 30-60 million dendritic cells on days 2, 8, and 15 of cycles 2 and 3, and day 2 of cycles 4 and 5. Patients undergo cryosurgery on day 2 of cycle 2 and receive pneumococcal 13-valent conjugate vaccine by injection on day 2 of cycles 2-5. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients who are CR, PR, or SD after completion of therapy, may receive pembrolizumab for an additional 18 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Started | 3 | 8
Completed | 3 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1 | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [56 to 79] | 64 [47.5 to 71] | 59 [56 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 8 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 8 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Experienced a Dose Limiting Toxicity (DLT)
Description: Maximum tolerated dose (MTD) will be defined as the dose level that does not induce dose limiting toxicity in at least one-third of patients. DLTs are defined as Grade 4 or 5 ANC or PLT for at least 7 days, grade 3 plus Infections and infestations, febrile neutropenia defined as fever ≥38.5oC (38 >1 hour) with grade 4 plus neutropenia, at least Grade 3 erythema multiforme, ulceration, or urticaria that does not resolve to Grade 2 or less within > three weeks, at least grade 3 bronchial obstruction, pneumonitis, or wheezing at least grade 3 allergic reaction or autoimmunity at least grade 3 that does not resolve to less than Grade 2> less than or equal to 72 hours per NCI Common Terminology Criteria for Adverse Events.
Time Frame: 56 days
Population: All eligible and treated phase 1 patients are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Percentage of Complete Responses of Combination Therapy With Pembrolizumab, Cryoablation, and Intra-tumor Injection of Autologous Dendritic Cells (DC) at Maximum Tolerated Dose (MTD) Dose
Description: The percentage of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated.
Time Frame: 24 months
Measure: Number; unit: percentage of patients
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Number analyzed (Participants) | 3 | 8
percentage of patients | 0 | 0

3. Secondary Outcome: Progression Free Survival
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Number analyzed (Participants) | 3 | 8
Months | 5 [3.8 to NA] — Not enough events occurred to calculate the upper confidence interval. | 3.6 [2.9 to NA] — Not enough events occurred to calculate the upper confidence interval.

4. Secondary Outcome: Treatment Free Survival
Description: The distribution of treatment-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: 34 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Number analyzed (Participants) | 1 | 3
months | 15.8 [NA to NA] — Not enough events to calculate the confidence interval. | 18.1 [5.2 to NA] — Not enough events to calculate the upper confidence interval.

5. Secondary Outcome: Duration of Response
Description: The distribution of duration of complete response will be estimated using the method of Kaplan-Meier.
Time Frame: 11 months
Population: Both phases were combined per protocol for this analysis. Only patients that achieved a response are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Patients: Patients receive 200mg pembrolizumab IV on day 1. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive an injection of between 30-60 million dendritic cells on days 2, 8, and 15 of cycles 2 and 3, and day 2 of cycles 4 and 5. Patients undergo cryosurgery on day 2 of cycle 2 and receive pneumococcal 13-valent conjugate vaccine by injection on day 2 of cycles 2-5. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients who are CR, PR, or SD after completion of therapy, may receive pembrolizumab for an additional 18 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Patients
Number analyzed (Participants) | 4
months | 6 [1.4 to NA] — Not enough events to calculate the upper confidence interval.

6. Secondary Outcome: Disease Free Survival Rate
Description: The percentage of patients without disease at two years post start of treatment.
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Number analyzed (Participants) | 3 | 8
percentage of patients | 0 | 0

7. Secondary Outcome: Overall Survival
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Number analyzed (Participants) | 3 | 8
months | NA [3.8 to NA] — Not enough events to calculate the median or upper confidence interval. | NA [3.6 to NA] — Not enough events to calculate the median or upper confidence interval.

8. Secondary Outcome: Percentage of Patients With Grade 4 or 5 Adverse Events
Description: Will be assessed by Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Number analyzed (Participants) | 3 | 8
percentage of patients | 0 | 0

9. Secondary Outcome: Percent of Patients With Improved Quality of Life
Description: Will be measured using the Functional Assessment of Cancer Therapy-lymphoma. The assessment will be scored according to the scoring algorithm. Changes from baseline will be calculated at each assessment time points. Mean change scores at each time point will be calculated to determine if quality of life is reduced over the course of treatment. Longitudinal techniques will be employed to describe changes over time.
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
Number analyzed (Participants) | 3 | 7
percentage of participants | 33.3 | 57.14

10. Other Pre Specified Outcome: Radiologic Analysis
Description: Measurements of index lesion(s) (non-cryoablated lesion) will be evaluated over time for each patient as a marker of systemic immune and treatment response to pembrolizumab and localized treatment with cryoablation and dendritic cell therapy. The index lesion(s) will be selected by the treating physician/investigator and are noncryoablated node. The percent change from baseline in index lesion measurements will be assessed over time. Differences in values over time will be summarized descriptively and graphically. The whole body computed tomography (CT) or positron emission tomography/CT will be used to assess overall clinical response and time to progression using the standard Cheson criteria.
Time Frame: Up to 4 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Immunologic Correlates
Description: Will be evaluated and summarized both quantitatively and graphically. Each of the correlative endpoints will be summarized individually, but will also be evaluated in terms of their relationships to one another; i.e., will use Spearman rank correlation coefficient to assess the correlations between baseline levels as well as between changes before and after treatment in these immunologic markers. In addition, these immunologic markers will be correlated with cancer and treatment- related outcomes (e.g. response, toxicities). Relationships will also be explored graphically using scatter plots.
Time Frame: Baseline up to 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events time frame was 4 years, mortality time frame was 5 years.
Arm/Group | Phase 1 Dose Level 1 | Phase 2 Dose Level 1
All-Cause Mortality (participants affected / at risk) | 1/3 | 4/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/8
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 2 Dose Level 1 (N=8)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 2 Dose Level 1 (N=8)
Anemia (Blood and lymphatic system disorders) | 2 (15) | 7 (39)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 5 (21)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (17)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (7)
Pain (General disorders) | 0 (0) | 2 (3)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (6)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (4)
Platelet count decreased (Investigations) | 1 (18) | 3 (7)
White blood cell decreased (Investigations) | 0 (0) | 1 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 2 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 2 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (16) | 4 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT03035331/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT03035331/ICF_001.pdf